CLINICAL TRIAL: NCT04065672
Title: Efficacy and Safety of Low-Dose Interleukin 2 for Behçet's Syndrome: a Phase 2, Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Low-dose IL-2 Treatment on Behcet's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HeJing (Other)
Responsible Party: Sponsor-Investigator, HeJing, professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019PHB089-03
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Behcet's Disease
Keywords: Behçet's syndrome; LD-IL-2 therapy; Treg cells; T follicular cells; Th17 cells
MeSH Terms: conditions — Behcet Syndrome | interventions — Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators and the study participants were masked to the allocation sequence and the intervention (study drug containing IL-2 or placebo). The study drug was packaged, labeled, and randomly assigned by an independent third party (Beijing Stemexel Technology Co).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose IL-2 (Experimental): After a 4-week screening period, patients received IL-2 at a dose of 1 million IU subcutaneously every other day. After the initiation of the therapy, patients could continue with concurrent medication but were prohibited from changing or adding immunosuppression therapy during the course of the study with a 12-week observational followed up.
  Interventions: Drug: Low-dose IL-2
- placebo (Placebo Comparator): After a 4-week screening period, patients received placebo subcutaneously every other day. After the initiation of the therapy, patients could continue with concurrent medication but were prohibited from changing or adding immunosuppression therapy during the course of the study with a 12-week observational followed up.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-dose IL-2 — After a 4-week screening period, patients received IL-2 at a dose of 1 million IU subcutaneously every other day. After the initiation of the therapy, patients could continue with concurrent medication but were prohibited from changing or adding immunosuppression therapy during the course of the study with a 12-week observational followed up.
  Arms: Low-dose IL-2
Drug: Placebo — After a 4-week screening period, patients received placebo subcutaneously every other day. After the initiation of the therapy, patients could continue with concurrent medication but were prohibited from changing or adding immunosuppression therapy during the course of the study with a 12-week observational followed up.
  Arms: placebo

SUMMARY:
The study aims to explore the clinical and immunological efficacy of low-dose IL-2 on Behcet's Disease.

DETAILED DESCRIPTION:
The investigators designed a single center, Phase 2, randomised, double-blind, placebo-controlled, parallel-group, superiority design study that routinely administered low-dose IL-2 therapy to monitor the improvement of clinical and laboratory parameters to explore its efficacy and to observe changes in immune cell subsets and cytokines. After a 4-week screening period, patients were randomly assigned in a 1:1 ratio to receive IL-2 at a dose of 1 million IU or placebo subcutaneously every other day. After the initiation of the therapy, patients could continue with concurrent medication but were prohibited from changing or adding immunosuppression therapy during the course of the study. After 12 weeks placebo-controlled treatment period, a 12-week observational followed up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-70 years of age at time of screening.
2. Diagnosis of Behçet's Disease (according to the 1989 ICBD) for ≥3 months before screening.
3. Active oral ulcer at time of screening.
4. Patients on corticosteroids (≤1 mg/kg/d prednisone or equivalent), DMARDs (e.g. methotrexate, hydroxychloroquine, azathioprine, MMF, leflunomide, ciclosporin etc.), must have been on a stable dose for 4 weeks prior to receiving the first infusion of study medication and expected to remain on this dose throughout the study. If the registered doctor plans to quit using current DMARDs or glucocorticoids, the washout period needs to be followed before patients join the groups. Each drug needs to meet the following washout period

   * glucocorticoids - 2 weeks
   * DMARDs (including mmethotrexate, hydroxychloroquine, azathioprine, MMF, leflunomide, and ciclosporin ) - 4 weeks
   * IVIg or cyclophosphamide - 2 months
   * Rituximab - 6 months
   * other bDMARDs(e.g. Infliximab, Adalimumab, Enanercept etc.) - 12 weeks
5. Given their written informed consent to participate in the trial and expected to be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. BD-related active major organ involvement requiring immunosuppressive therapy, e.g., pulmonary (e.g., pulmonary artery aneurysm), vascular (e.g., thrombophlebitis, recurrent malignant aneurysms), gastrointestinal (e.g., gastrointestinal ulcers), and central nervous system (e.g., meningoencephalitis).
2. High-dose glucocorticoid (>1mg/kg/d) usage within 1 month.
3. Severe comorbidities: including Heart failure (≥ grade III NYHA); Renal insufficiency (creatinine clearance ≤30 ml/min); Hepatic insufficiency (serum ALT or AST >3 times the ULN, or total bilirubin >ULN for the central laboratory conducting the test).
4. Other severe, progressive or uncontrolled hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease (including demyelinating diseases such as multiple sclerosis).
5. Known allergies, hypersensitivity, or intolerance to IL-2 or its excipients.
6. History of severe allergic reaction to monoclonal antibodies or to murine, chimeric, or human proteins or their excipients.
7. Had a severe infection (including, but not limited to hepatitis, pneumonia, sepsis, or pyelonephritis); had been hospitalized for an infection; or had been treated with IV antibiotics for an infection, within 2 months prior to the first administration of study agent.
8. Chest radiograph within 3 months prior to the first administration of study agent that showed an abnormality suggestive of a malignancy or current active infection, including TB.
9. Infected with HIV (positive serology for HIV antibody) or hepatitis C (positive serology for Hep C antibody). If seropositive, consultation with a physician with expertise in the treatment of HIV or hepatitis C virus infection was recommended.
10. Infected with hepatitis B virus. For patients who were not eligible for this study due to hepatitis B virus test results, consultation with a physician with expertise in the treatment of hepatitis B virus infection was recommended.
11. Had any known malignancy or has a history of malignancy within the previous 5 years (with the exception of a nonmelanoma skin cancer that had been treated with no evidence of recurrence for ≥3 months before the first study agent administration or cervical neoplasia with surgical cure).
12. Had uncontrolled psychiatric or emotional disorder, including a history of drug and alcohol abuse within the past 3 years that might prevent the successful completion of the study.
13. Received, or was expected to receive, any live virus or bacterial vaccination within 3 months before the first administration of study agent, during the study, or within 4 months after the last administration of study agent. Had a BCG vaccination within 12 months of screening.
14. Pregnancy, lactation or women of child-bearing potential (WCBP) unwilling to use medically approved contraception whilst receiving treatment and for 12 months after treatment has finished.
15. Men whose partners are of child-bearing potential but who are unwilling to use appropriate medically approved contraception whilst receiving treatment and for 12 months after treatment has finished.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
the number of oral ulcers at week 12 | Week 12
  the number of oral ulcers at week 12

SECONDARY OUTCOMES:
the change in pain from oral ulcers from baseline to week 12 | Week 12 and Week 24
  measured on a 100-mm visual-analogue scale (with 0 representing nopain and 100 the worst pain ever experienced),and the change in disease activity from baselineto week 12.
Change from baseline in the Behçet's Syndrome Activity Score | Week 12 and Week 24
  a scaleon which scores range from 0 to 100, with higherscores indicating more active disease
Change from baseline in simplified Behcet Disease Current Activity Form (BDCAF) Score | Week 12 and Week 24
  cores range from 0 to 12, withhigher scores indicating more active disease
Change from baseline in Protocol-specific immunophenotypic analysis of peripheral blood lymphocyte subsets | Week 12 and Week 24
  Relative proportions of Treg, Tfh, Th1, Th2 and Th17 cell subsets were analyzed by flow cytometetry usingFACSAria III (BD) and FlowJo software (Tree Star). Treg cells were defined as CD3+ CD4+ CD25high CD127low, Tfh cells as CD3+ CD4+ CXCR5+ PD1high CCR7low6, Th1 cells as CD3+ CD4+ CXCR3+ CCR6- CCR4- CCR7low, Th2 cells as CD3+ CD4+ CXCR3+ CCR6- CCR4+ CCR7low and Th17 cells as CD3+ CD4+ CXCR3- CCR6+ CCR4+ CCR7low26.
the number of genital ulcers at week 12 and Week 24 | Week 12 and Week 24
  the number of genital ulcers at week 12 and Week 24
the proportion of patients with a complete response to oral ulcers | Week 12
  the proportion of patients who had no oral ulcers at week 12
the percentage of patients with genital ulcers at baseline who were ulcer-free at week 12 | Week 12
  the percentage of patients with genital ulcers at baseline who were ulcer-free at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, MD,PhD, Principal Investigator — Department of Rheumatology and Immunology, Peking University People's Hospital.
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunduz E, Teke HU, Bilge NS, Cansu DU, Bal C, Korkmaz C, Gulbas Z. Regulatory T cells in Behcet's disease: is there a correlation with disease activity? Does regulatory T cell type matter? Rheumatol Int. 2013 Dec;33(12):3049-54. doi: 10.1007/s00296-013-2835-8. Epub 2013 Aug 3. PMID 23912800
- [Background] Nanke Y, Kotake S, Goto M, Ujihara H, Matsubara M, Kamatani N. Decreased percentages of regulatory T cells in peripheral blood of patients with Behcet's disease before ocular attack: a possible predictive marker of ocular attack. Mod Rheumatol. 2008;18(4):354-8. doi: 10.1007/s10165-008-0064-x. Epub 2008 Apr 22. PMID 18427720
- [Background] Mohammadi M, Shahram F, Shams H, Akhlaghi M, Ashofteh F, Davatchi F. High-dose intravenous steroid pulse therapy in ocular involvement of Behcet's disease: a pilot double-blind controlled study. Int J Rheum Dis. 2017 Sep;20(9):1269-1276. doi: 10.1111/1756-185X.13095. Epub 2017 May 19. PMID 28524639
- [Background] Zou J, Ji DN, Shen Y, Guan JL, Zheng SB. Mucosal Healing at 14 Weeks Predicts better Outcome in Low-dose Infliximab Treatment for Chinese Patients with Active Intestinal Behcet's Disease. Ann Clin Lab Sci. 2017 Mar;47(2):171-177. PMID 28442519
- See also: Primary outcome for BD patients — http://www.clinicaltrials.gov